CLINICAL TRIAL: NCT04642846
Title: Clinical and Laboratory Assessments of Effectiveness of Silver Diamine Fluoride (SDF) in Arresting Caries Among Children and Parental ￼Satisfaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khalood Saeed Bahammam (Other)
Responsible Party: Sponsor-Investigator, Khalood Saeed Bahammam, Intern at Imam Abdulrahman Bin Faisal University, Imam Abdulrahman Bin Faisal University
Organization: Imam Abdulrahman Bin Faisal University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IAU
Record Dates: First submitted 2020-10-07; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Caries Arrested
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- one application of SDF (Experimental)
  Interventions: Other: Silver Diamine Fluoride (SDF)
- two application of SDF one month apart (Experimental)
  Interventions: Other: Silver Diamine Fluoride (SDF)

INTERVENTIONS:
Other: Silver Diamine Fluoride (SDF) — Silver diamine fluoride (SDF) is one of the topical methods for caries arresting. The advantages of using SDF include ease of use, low cost, pain and infection control, minimal requirement of time/training and non-invasive nature of the procedure. SDF can improve oral health, increase access to care and reduce the need for emergency treatment

SUMMARY:
Globally, it is estimated that 2.4 billion people suffer from caries of permanent teeth and 486 million children suffer from caries of primary teeth . The highest estimate of dental caries prevalence in Saudi Arabia was 95% with maximum DMFT of 7.34 among 3-7 years old children . Also, it was found that 78% of 6-9 years old children in Dammam had caries with an average of 3.66±3.13 DMFT.

The objectives of this study are:

1. To assess the effectiveness of the Silver Diamine Fluoride (SDF) in arresting caries.
2. To assess the antibacterial effect of the Silver Diamine Fluoride (SDF).
3. To assess parents' and children's satisfaction and acceptance.

The aims of our study are to assess the effectiveness of SDF in arresting caries in primary dentition among children visiting Imam Abdulrahman bin Faisal University in Dammam, Saudi Arabia and to assess parental acceptance and satisfaction.

The expected outcome the results of this study will help in understanding the effectiveness SDF in arresting dental caries in this target population especially that it was recently approved for clinical use in Saudi Arabia.

ELIGIBILITY:
Inclusion Criteria:

* Children between four and six years of age.
* Healthy.
* Have at least two active dentin carious lesions on the primary teeth meeting the International Caries Detection and Assessment System (ICDAS) score 5 or 6.
* Should not have periapical infection, root resorption or widening in the periodontal ligament space.

Exclusion Criteria:

* Participants who have systemic or neurological diseases.
* Tooth abscess, pain on percussion, symptoms of pulpal involvement or mobility,
* Allergic to silver or any dental material to be used.
* Unable to attend follow-up visits.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 155 (Estimated)
Dates: Start 2020-11-21 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the Silver Diamine Fluoride (SDF) in arresting caries. | 2 years
  Caries arresting rate: total number of arrested teeth/ total number of treated teeth.

SECONDARY OUTCOMES:
Clinical changes of dentinal lesion: in the hardness and softness. | 2 years
  Changes in ICDAS score: post treatment change in carious lesion status.
The antibacterial effect of the Silver Diamine Fluoride (SDF). | 2 years
  by DNA extractions and performed the 16S rRNA sequencing
Parents satisfaction | 2 years
  To assess parents' and children's satisfaction and acceptance by questionnaire (Arabic and English). Link: https://forms.office.com/Pages/ResponsePage.aspx?id=_LuGLASN_0GoOpQvB14PYCVJ8_tHLjNCkOqqrov3N-1UMFlYRzFQUVRKMDhNUEtJR1ZXNkk4SzhGWS4u

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Abdulrahman Bin Faisal University, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided